CLINICAL TRIAL: NCT06540092
Title: Early Pregnancy Ultrasound Measurements and Prediction of First Trimester Pregnancy Loss.
Status: Completed | Type: Observational
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Hend Mahmoud Abdelghany, Lecturer of Obstetrics and Gynecology, Cairo University, Kasr El Aini Hospital
Other Study IDs: MS-521-2023
Record Dates: First submitted 2024-08-01; First posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: First Trimester Abortion
Keywords: ultrasound measurments
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: ultrasound — ultrasound measurements during first trimester

SUMMARY:
Ultrasound measurements of fetus during first trimester may be an indicator of first trimester pregnancy loss. Investigators took 4 measurements of the fetus on 2 intervals during first trimester to confirm this hypothesis.

DETAILED DESCRIPTION:
Ultrasound examination of gestational sac (GS) diameter, yolk sac (YS) diameter, crown rump length (CRL) diameter, embryonal heart rate (HR) using Samsung Medison SonoAce R3 through transvaginal probes (6.5 MHz) was conducted on 126 pregnant women. At least 2 scans were done for each participant one between 6-8 weeks and another one by the end of first trimester. Results then were compared to get the cut off values that can predict pregnancy loss.

ELIGIBILITY:
Inclusion Criteria:

* • Healthy pregnant female patient in the reproductive age group; 18 - 40 years old.

  * Gestational age: 6 - 13 weeks of gestations.
  * Singlton or multifetal pregnancy.
  * Any mode of conception included spontaneous, after superovulation with clomiphene citrate or letrozole with, or without, intrauterine insemination (IUI), and in vitro fertilization (IVF) after superovulation with gonadotropins.

Exclusion Criteria:

* • Patient with unsure date for the last menstrual period.

  * Pregnant women above 13 weeks gestation.
  * Patient with symptoms of threatened abortion or ectopic pregnancy at the initial antenatal visit.
  * Patient unable to come for follow up.
  * Any medical disorders as DM, HTN, …

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 126 pregnant women between 6- 13 weeks
Sampling Method: Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2024-03-19 (Actual); Primary Completion 2024-06-26 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
The relation between early pregnancy ultrasound measurements (GSD, YSD, CRL, HR), viability, and continuation of pregnancy till 13 weeks of gestation. | 6-7 weeks
  2 measures of the fetus were obtained and compared to get first trimester pregnancy outcome

CONTACTS AND LOCATIONS:
Locations (1):
- kasr Al Aini, Faculty of Medicine, Cairo University, Cairo, Old Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No